CLINICAL TRIAL: NCT00549263
Title: A Bioequivalence Study With a Combination Tablet Formulation of Rosiglitazone (RSG) and Glimepiride (GLIM)(4mg/2mg) Compared to Concomitant Dosing of RSG 4mg Tablet and GLIM 1mg Commercial Tablet x 2 (4mg+2mg) in Japanese Healthy Male Subjects
Brief Title: Bioequivalence Study of SB797620 in Healthy Japanese Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No subjects enrolled, bio equivalence study, canceled before active.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AVR110549
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Subjects
Keywords: Safety; Pharmacokinetics; Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB797620

SUMMARY:
This study will test whether the Drug levels in plasma after combination formulation tablet dosing (SB797620) and separate formulation tablets dosing (rosiglitazone and glimepiride) to Japanese Healthy volunteer would be the same or not.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* They are Japanese males.
* Aged 20 to 55 years, inclusive.
* They have body mass index at screening within 18.5-25.0. Body weight 50-80kg.
* AST(GOT), ALT(GPT), gumma-GPT and ALP: below the upper normal range
* They are capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* They could refrain from smoking during hospitalization.
* They are able to attend all visits and complete the study.

Exclusion Criteria:

* The subject has any clinically relevant abnormality on medical examination, vital sign, clinical laboratory test or medical history at screening in the medical opinion of the investigator or the subject has a medical history that is not considered as eligible for inclusion in this study by the investigator.
* Known hepatic or biliary abnormalities such as Gilbert's syndrome.
* Use of insulin or oral anti-hyperglycemic agents within the past 3 months prior to screening.
* Subjects who have a history of lactose intolerance.
* The subject has an allergy for any drug or idiosyncrasy. This excludes a pollen allergy without current symptoms.
* The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* The subject has participated in a clinical study with an investigational or a non-investigational drug or device during the previous 4 months.
* The subject has a screening ECG with a QTc value outside the range 320 to 450msec, a PR interval of >230msec and/or a QRS interval of >120msec.
* The subject has a heart rate outside the range 40 to 110 bpm at screening.
* The subject has donated a unit of blood ">400mL" within the previous 4 months or ">200mL" within the previous 1 month.
* The subject is currently taking regular (or a course of) medication (including prescribed drug, over-the-counter medication and herbal remedies), and can not cease them 30 days prior to th first study drug dosing.
* The subject has a history or current conditions of drug abuse or alcoholism.
* History of alcohol consumption in the past six months exceeding 7 drinks per week (where 1 drink is 350mL in terms of beer)
* The subject is positive for syphilis, HBs antigen, HCV antibody, HIV antigen/antibody, HTLV-1 antibody.
* The subject is positive for urine drug screening.
* Current history of hypo- or hyperglycemia as indicated by serum glucose values below the laboratory-specified reference range or =110 mg/dL, at screening, or as reported by the subject.
* History of surgical procedures that might affect the absorption of RSG or GLIM (e.g., partial/total gastrectomy, cholecystectomy).
* History of hypersensitivity to thiazolidinediones, sulfonylureas or compounds with similar chemical structures.
* History of sensitivity to heparin, heparin-induced thrombocytopenia or sensitivity to any of the study medications or components thereof.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Drug levels on Day 1 | Day 1

SECONDARY OUTCOMES:
Adverse events on Day 1 | Day 1
Clinical laboratory test on Day 1 | Day 1
Vital signs and 12-lead ECG on Day 1 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline